CLINICAL TRIAL: NCT06254365
Title: Effects of Antagonizing the Ghrelin Receptor on Total-body Glucose Metabolism in Obesity
Brief Title: Investigating Glucose Metabolism of LEAP2 With Total-body PET/CT
Acronym: LEAP2-PET/CT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, MD, PhD, Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: H-23042551; NNF20OC0084114 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2024-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LEAP2 infusion then placebo infusion (Experimental): Participants are randomized to either first recieve LEAP2 infusion and then LEAP2 infusion or th other way around.
  This arm describes - first LEAP2 infusion and then placebo infusion
  Interventions: Biological: Exogenous LEAP2 hormone
- Placebo infusion then LEAP2 infusion (Experimental): Participants are randomized to either first recieve LEAP2 infusion and then LEAP2 infusion or th other way around.
  This arm describes - first placebo infusion and then LEAP2 infusion
  Interventions: Biological: Exogenous LEAP2 hormone

INTERVENTIONS:
Biological: Exogenous LEAP2 hormone — This intervention has never been examined in this type of study before.

SUMMARY:
The naturally occurring hormone LEAP2 is proposed to have opposite effects to that of the 'hunger hormone' ghrelin. Other that appetite regulation, LEAP2 is involved in glucose metabolism through mechanisms yet not fully understood. With two experimental days; one recieving LEAP2 and one recieving placebo infusion in a randomized order, the study will explore the effect of LEAP2 (vs. placebo) on glucose metabolism through total-body PET/CT-scans and thereby gain a deeper understanding of the ghrelin/LEAP2 system and its interaction with glucose metabolism. Furthermore, the project will generate scanning references in individuals with obesity that are usable in forthcoming research projects.

DETAILED DESCRIPTION:
Regulation of appetite and glucose metabolism involves complex and partially unknown mechanisms; it is however well-established that the gastric hormone ghrelin increases appetite through the central nervous system and increases plasma glucose levels through various organs and tissues. The role of ghrelin has been investigated in diseases and conditions with dysregulated appetite control such as anorexia nervosa and obesity but the full picture of ghrelin receptor signalling remains unclear. Despite recent advances in medical therapies for obesity management, bariatric surgery is the most effective treatment for severe obesity and related complications . The weight-reducing and beneficial metabolic effects of the most used bariatric procedures relies mainly on changes in appetite-regulating gut hormones after the operation. Center for Clinical Metabolic Research have previously examined the molecular phenotype of enteroendocrine cells in the small intestine following the bariatric surgical procedure Roux-en-Y gastric bypass (RYGB) in individuals with obesity with and without type 2 diabetes. Through transcriptomics, Center for Clinical Metabolic Research discovered that the gene encoding liver enriched antimicrobial peptide 2 (LEAP2), a naturally occurring human peptide, was significantly upregulated compared to baseline expression. LEAP2 is a competitive antagonist/inverse agonist of the ghrelin receptor counteracting ghrelin-induced food intake in mice and LEAP2 may contribute to our understanding of appetite and gluco-metabolic alterations going through the ghrelin recepto. In recent studies, Center for Clinical Metabolic Research have found that ghrelin receptor-antagonism/infusion of LEAP2 improves postprandial glucose tolerance and decreases ad libitum food intake in both healthy, lean individuals and individuals with obesity compared to placebo. However, the mechanisms involved in reduced preprandial and postprandial glucose responses during ghrelin receptor-antagonism remain unclear.

Positron emission tomography (PET) is a functional imaging technique that uses radioactively labelled tracers to visualize physiology, including perfusion and metabolism. When the radioactive isotope undergo decay, it emits a positron, which travels a few millimetres in the tissue and collides with an electron, the two particles annihilate, and two photons are emitted in opposite directions. The photons hit detectors and are, thus, registered, and the detected data can then be transformed into images. In the present study the investigators will use the most frequently used PET tracer 18F-fluoro-deoxy-glucose (FDG), which is a glucose analogue. The molecular structure of FDG is very similar to that of glucose, and the tracer is, therefore, expected to be an appropriate representative for glucose metabolism. Today, PET is combined with computed tomography (CT) to form an anatomical foundation for the scan. CT scans use X-rays to create detailed cross-sectional images of the body's various tissues and organs. Conventional PET systems typically have a 20-25 cm axial field of view (FOV) and they are primarily used as a tool for examining cancer, infection and inflammatory diseases. In 2021, a Siemens Vision Quadra total-body PET-CT scanner (Quadra) was installed at Copenhagen University Hospital (Rigshospitalet) as one of the first of its kind in Europe. The Quadra has a long axial FOV of 106 cm and it can, thus, acquire dynamic data from all major organs, including the brain, in only one bed position. The Quadra has up to 40 times higher sensitivity than previous PET-CT scanners, and further, scans can be made much faster and/or with lower radiation doses without deterioration of image quality . The long FOV enables quantitation of tracer uptake in all organs simultaneously, which means that the interplay between different organs systems (e.g. the gut-brain axis) now can be visualized, which has not been possible before. Furthermore, due to the high temporal resolution of total-body PET, it is possible to quantitate organ perfusion with all PET tracers. Finally, the increased sensitivity enables detection of even minor changes in organ perfusion and metabolism.

Our overall objective is to investigate the effects of the naturally occurring ghrelin receptor antagonist on human glucose metabolism using innovative total-body PET-CT based techniques. The study will explore the effect of exogenous LEAP2 (vs. placebo) on dynamic FDG uptake and thereby examine uptake rates and biodistribution of glucose to gain a deeper understanding of the ghrelin system and its interaction with glucose metabolism. Furthermore, the project will generate reference FDG total-body PET data in obese individuals that are usable in forthcoming research projects.

The study is a randomized, placebo-controlled, single-blind crossover study comprising two experimental days for each participant with intravenous (i.v.) infusion of LEAP2 and placebo, respectively. On experimental days, participants will undergo a total-body PET/CT scan preceded by i.v. administration of FDG. PET/CT measurements of dynamic FDG uptake and distribution will be recorded for 70 min following administration of FDG. A low dose CT combined with in-house developed deep-learning algorithm will be applied for attenuation correction. Nine individuals with obesity will be included.

Primary outcome:

Ghrelin increases plasma levels of glucose and, therefore, the investigators hypothesise that the ghrelin receptor antagonist will increase the metabolic rate of glucose (MRglu) in organs of interest assessed with total-body PET/CT scans compared to placebo (saline) in individuals with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Age between 18 and 60 years at the time of inclusion
* Body mass index 30-50 kg/m2
* Informed consent

Exclusion Criteria:

* Anaemia (haemoglobin below normal range)
* Alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) ≥2 times normal values) or present hepatobiliary and/or gastrointestinal disorder(s)
* Nephropathy (serum creatinine above normal range and/or albuminuria)
* Glycated haemoglobin (HbA1c) ≥48 mmol/mol and/or type 2 diabetes requiring medical treatment
* Regular tobacco smoking or use of other nicotine-containing products
* Claustrophobia
* Any ongoing medication that the investigator evaluates would interfere with trial participation.
* Any physical or psychological condition that the investigator evaluates would interfere with trial participation including any acute or chronic illnesses

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 9 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in in hepatic MRglu (metabolic rate of glucose) | During PET-scan (From time 75 minutes to 145 minutes)
  The primary endpoint is the change in hepatic MRglu (metabolic rate of glucose) assessed with total-body PET/CT technique, which will be compared between the two experimental days with infusion of placebo and LEAP2, respectively

SECONDARY OUTCOMES:
Standardized uptake values (SUVs) | During PET-scan (From time 75 minutes to 145 minutes)
  Mean and maximum standardized uptake values (SUVs) in organs of interest
Change MRglu (metabolic rate of glucose) in organs of interest | During PET-scan (From time 75 minutes to 145 minutes)
  MRglu in other organs of interest
Hepatic intracellular phosphorylation rate | During PET-scan (From time 75 minutes to 145 minutes)
  Hepatic intracellular phosphorylation rate of glucose
Hepatic glucose influx and efflux rates | During PET-scan (From time 75 minutes to 145 minutes)
  Hepatic glucose influx and efflux rates
Plasma glucose | During PET-scan (From time 75 minutes to 145 minutes)
  Plasma glucose levels
LEAP2 levels | During entire experimental day (From time -15 minutes to 145 minutes)
  LEAP2 levels
Growth hormone levels | During entire experimental day (From time -15 minutes to 145 minutes)
  Growth hormone levels
Insulin levels | During entire experimental day (From time -15 minutes to 145 minutes)
  Insulin levels
C-peptide levels | During entire experimental day (From time -15 minutes to 145 minutes)
  C-peptide levels

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Professor, Principal Investigator — Center for Clinical Metabolic Research, Gentofte Hospital
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No